CLINICAL TRIAL: NCT06936683
Title: Prognostic Effect of Herpes Simplex Virus Type 1 Infection/Reactivation in the Lower Respiratory Tract of Critical Care Patients With Severe Pneumonia（the HSV-SP Study）: a Study Protocol for a Multicenter, Prospective Cohort Study
Brief Title: Herpes Simplex Virus Type 1 Infection/Reactivation of Patients With Severe Pneumonia（the HSV-SP Study）
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Guangzhou Red Cross Hospital (Other); Guangzhou First People's Hospital (Other); Gongguan People's Hospital (Unknown); Guangzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: MR-44-24-013041
Record Dates: First submitted 2025-04-14; First posted 2025-04-20 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Severe Pneumonia
Keywords: Severe pneumonia; Herpes simplex virus type 1; infection/reactivation; Prognostic effect
MeSH Terms: conditions — Pneumonia; Latent Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage fluid (BALF) is a sterile saline solution collected from the lungs during a procedure called bronchoalveolar lavage. A thin, flexible tube (bronchoscope) is inserted into the airways, and saline is gently instilled into a specific lung segment. The fluid is then suctioned back, carrying cells, proteins, and microorganisms from the alveoli (tiny air sacs).
  BALF is analyzed to diagnose lung infections (e.g., pneumonia), inflammatory diseases (e.g., sarcoidosis), or cancers. It provides critical information about immune cells, pathogens, and biomarkers in the lower respiratory tract.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Bronchoalveolar Lavage (BAL) via Fiberoptic Bronchoscopy — Bronchoalveolar Lavage (BAL) via Fiberoptic Bronchoscopy
  1. Site selection: For patients with limited lesions, the lesion segment was chosen; For patients with diffuse lesions, the right middle lobe or left upper lobe tongue should be severed.
  2. Injecting physiological saline: After the top of the bronchoscope is embedded in the target bronchial segment or subsegment opening, 37 ℃ or room temperature physiological saline is rapidly injected through the operating channel, with a total volume of 60-120ml, injected in batches (20-50ml each time).
  3. Negative pressure suction: After injecting physiological saline, immediately use appropriate negative pressure (generally recommended below 100mmHg) to suction and obtain BALF, with a total recovery rate of ≥ 30%.
  4. BALF collection: Specimens used for pathogen analysis need to be collected in sterile containers; Cytological analysis requires the selection of plastic containers or siliconized glass containers to reduce cell adhesion.
Diagnostic Test: throat Swab — A throat swab is a diagnostic sampling technique used to collect microbial specimens from the oropharynx and tonsillar areas. The standardized procedure involves:
  1. Positioning the patient with their head tilted slightly backward;
  2. Using a sterile, synthetic-fiber swab with a plastic shaft (avoiding calcium alginate or wooden shafts);
  3. Vigorously rubbing the swab over both tonsillar pillars and the posterior pharyngeal wall while avoiding contact with the tongue, teeth, or uvula;
  4. Immediately placing the swab into appropriate transport media viral/bacterial);
  5. Maintaining cold chain (2-8°C) for specimen transport if required.

SUMMARY:
Severe pneumonia(SP) is a one of the main causes of death for critically ill patients.Samples of bronchoalveolar lavage fluid (BALF) from SP patients often report positive for herpes simplex virus type 1 (HSV-1) DNA. However, to date, it is unclear the impact and significance of this positive result on SP patients. This study will evaluate the prognostic impact of lower respiratory tract HSV-1 infection/reactivation on ICU severe pneumonia patients.At the same time, by analyzing the risk factors that affect prognosis, we will identify populations with the potential for intervention benefits and provide a basis for further intervention treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1: Age>18 years old. 2: Clinical diagnosis for severe pneumonia. 3: ICU stay time >72 hours. 4: A written informed consent form was obtained from the members of the patients' family.

Exclusion Criteria:

* 1: severe ventilation dysfunction, and effective respiratory support has not been used; 2: Aortic aneurysm and esophageal varices at risk of rupture; 3: Recent acute coronary syndrome, uncontrolled severe hypertension, and malignant arrhythmia; 4: Irreversible bleeding tendencies, such as severe coagulation dysfunction, massive hemoptysis, or gastrointestinal bleeding; 5: Multiple pulmonary bullae at risk of rupture. 6: Estimated survival time<24 hours. 7: Included in another interventional clinical study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population Description ：Patients with age>18 years old admitted to the ICU who meet the diagnostic criteria for severe pneumonia.
Sampling Method: Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
30 day mortality rate of critical care patients with severe pneumonia. | From enrollment (Day 1) through Day 30

SECONDARY OUTCOMES:
The incidence rate of herpes simplex virus type 1 infection/reactivation in the lower respiratory tract of critical care patients with severe pneumonia | From enrollment (Day 1) through Day 30
ICU mortality and in-hospital mortality , ICU stay time and length of in-hospital stay | From enrollment (Day 1) through the entire ICU stays and in-hospital stays
success rate of ventilator withdrawal, ICU non ventilator survival time | From enrollment (Day 1) through Day 30